CLINICAL TRIAL: NCT00922480
Title: A Randomized, Double-blind, Losartan-controlled, Parallel Group Comparison Dose Titration Clinical Study to Evaluate the Antihypertensive Efficacy and Safety of Fimasartan 60mg~120mg in Patients With Mild to Moderate Essential Hypertension
Brief Title: Clinical Study to Evaluate the Antihypertensive Efficacy and Safety of Fimasartan in Hypertension Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Collaborators: Seoul National University Hospital (Other); The Catholic University of Korea (Other); Kangbuk Samsung Hospital (Other); Konkuk University Medical Center (Other); Konyang University Hospital (Other); Keimyung University (Other); Korea University (Other); Korea University Guro Hospital (Other); Dongguk University International Hospital (Other); Seoul National University Bundang Hospital (Other); Samsung Medical Center (Other); Asan Medical Center (Other); Severance Hospital (Other); Ajou University (Other); Wonju Severance Christian Hospital (Other); Yeungnam University Hospital (Other); Yonsei University (Other); Inha University Hospital (Other); Chonbuk National University Hospital (Other); Cheil General Hospital and Women's Healthcare Center (Other); Chungnam National University (Other); Chungbuk National University Hospital (Other); Hanyang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A657-BR-CT-301
Record Dates: First submitted 2009-06-16; First posted 2009-06-17 (Estimated); Results first posted 2018-02-13 (Actual); Last update posted 2018-04-10 (Actual); Status verified 2018-03

CONDITIONS: Hypertension
Keywords: Hypertension; Losartan
MeSH Terms: conditions — Hypertension | interventions — fimasartan; Losartan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2 (Active Comparator): Losartan group
  Interventions: Drug: Losartan (Control)
- 1 (Active Comparator): Fimasartan 60mg, 120mg
  Interventions: Drug: Fimasartan

INTERVENTIONS:
Drug: Fimasartan — Fimasartan 60 ~ 120mg/po take one tablets once a day
  Other Names: A657-BR-CT
  Arms: 1
Drug: Losartan (Control) — Losartan 50 mg ~ 100 mg/po, take one tablets once a day
  Other Names: Cozar
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the antihypertensive efficacy and safety of Fimasartan (BR-A-657•K) 60 mg~120 mg in patients with mild to moderate essential hypertension.

DETAILED DESCRIPTION:
Fimasartan (BR-A-657-K), a selective blocker of AT1 receptor subtype, showed the rapid and potent antihypertensive effect in many hypertensive models. Phase I study, Fimasartan (BR-A-657-K) 20mg ~ 480mg single dosing with healthy subjects, demonstrated that the Fimasartan(BR-A-657-K) was very safe and well tolerated. Another phase I study, Fimasartan (BR-A-657-K) 120mg and 360mg dosing for 7 days, also showed that Fimasartan (BR-A-657-K) was safe and tolerable though one temporal adverse event was observed in high dose.

A Randomized, Double-blind, Losartan-controlled, Parallel Group Comparison Dose Titration Clinical Study to Evaluate the Antihypertensive Efficacy and Safety of Fimasartan (BR-A-657•K) 60mg~120mg in Patients with Mild to Moderate Essential Hypertension.

Approximately 480 patients will be enrolled over 12 months in 24 centers nationwide.

After 2 weeks of placebo run-in period, all subjects will be randomized into one of the following 2 groups. Subjects will take test/control drug for 12 weeks of treatment period. And Extensin study have 12 weeks in treatment period.

If subjects take any antihypertensive medications before screening, the subjects will have 1 week of wash-out period.

If the hypertension is not controlled well, there is a possibility of dose titration.

Group I : Fimasartan group. Group II : Losartan group

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderate essential hypertension : sitting diastolic blood pressure measured at Placebo visit and Baseline are 90~109mmHg inclusive and the difference between sitting diastolic blood pressures measured at Placebo visit and Baseline(Day0) is under 7mmHg.
* Subjects who agree to participate in this sudy and give written informed consent
* Subjects considered to understand the study, be cooperative, and able to be followed-up until the end of the study

Exclusion Criteria:

* The sitting DBP is less than 89mmHg or more than 110mmHg or severe hypertensive patient with sitting systolic blood pressure over 200mmHg Patients with secondary hypertension
* Patients with severe renal(Creatinine more 1.5 times than upper limit of normal), gastrointestinal, hematological or hepatic(AST, ALT more 2 twice more than upper limit of normal)disease etc. which might affect absorption, disposition, metabolism or excretion of the drug
* Patients with postural hypotension
* Patients with sever insulin dependent diabetes mellitus or uncontrolled diabetes mellitus(HbA1c>9%, regimen change of oral hypoglycemic agents within 12weeks, treated insulin before screening)
* Patients with a history of myocardial infarction, severe coronary artery disease or clinically significant heart failure or valvular defect in last 6 months
* Patients with consumptive disease, autoimmune disease, connective tissue disease
* Patients with a history of type B or C hepatitis(include carrier)
* Patients with HIV or hepatitis
* Patients with clinically significant laboratory abnormality
* Patients receiving any drugs known to affect blood pressure or medical treatments that can influence the blood pressure
* Patients with allergy or contraindication to any angiotensin II receptor antagonists
* Female of childbearing potential who does not undergo hysterectomy or is not post-menopausal
* Patients judged to have a history of alcohol or drug abuse by the investigator
* Patients participated other clinical trial 12 weeks before Screening Patients judged to be inappropriate for this study by the investigator with other reasons

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 506 (Actual)
Dates: Start 2008-12; Primary Completion 2009-07 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Byung-Hee Oh, MD, Principal Investigator — Seoul National University Hospital

REFERENCES:
- [Derived] Lee SE, Kim YJ, Lee HY, Yang HM, Park CG, Kim JJ, Kim SK, Rhee MY, Oh BH; Investigators. Efficacy and tolerability of fimasartan, a new angiotensin receptor blocker, compared with losartan (50/100 mg): a 12-week, phase III, multicenter, prospective, randomized, double-blind, parallel-group, dose escalation clinical trial with an optional 12-week extension phase in adult Korean patients with mild-to-moderate hypertension. Clin Ther. 2012 Mar;34(3):552-568, 568.e1-9. doi: 10.1016/j.clinthera.2012.01.024. Epub 2012 Mar 3. PMID 22381711
- [Derived] Fimasartan. Am J Cardiovasc Drugs. 2011 Aug 1;11(4):249-52. doi: 10.2165/11533640-000000000-00000. PMID 21740078

RESULTS

PARTICIPANT FLOW:
Groups:
- Control: Losartan: Losartan group
  Losartan (Control): Losartan 50 mg ~ 100 mg/po, take one tablets once a day
- Test: Fimasartan: Fimasartan 60mg, 120mg
  Fimasartan: Fimasartan 60 ~ 120mg/po take one tablets once a day
Period: Main Study
Arm/Group | Control: Losartan | Test: Fimasartan
Started | 250 | 255
Completed | 213 | 226
Not Completed | 37 | 29
Not completed — Protocol Violation | 3 | 6
Not completed — Adverse Event | 6 | 7
Not completed — Lack of Efficacy | 3 | 0
Not completed — Withdrawal by Subject | 20 | 15
Not completed — Lost to Follow-up | 5 | 0
Not completed — Physician Decision | 0 | 1
Period: Extension Study
Arm/Group | Control: Losartan | Test: Fimasartan
Started | 73 | 85
Completed | 68 | 82
Not Completed | 5 | 3
Not completed — Protocol Violation | 3 | 0
Not completed — Adverse Event | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Others | 0 | 1

BASELINE CHARACTERISTICS:
Population: As ITT group, these are subjects who have been randomly assigned and have at least one primary end point.
Groups:
- Total: Total of all reporting groups
Arm/Group | Control: Losartan | Test: Fimasartan | Total
Number analyzed (Participants) | 238 | 247 | 485
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.58 (9.61) | 53.96 (8.79) | 53.77 (9.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71 | 79 | 150
  Male | 167 | 168 | 335

OUTCOME MEASURES:

1. Primary Outcome: Diastolic Blood Pressure Change
Description: Value of DBP at 12 Weeks minus value of DBP at Baseline while in a sitting position
Time Frame: baseline and 12 weeks
Population: As ITT group, these are subjects who have been randomly assigned and have at least one primary end point.
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Control: Losartan / Week 12 -ITT: Losartan group
  Losartan (Control): Losartan 50 mg ~ 100 mg/po, take one tablets once a day
- Test: Fimasartan / Week 12 -ITT: Fimasartan 60mg, 120mg
  Fimasartan: Fimasartan 60 ~ 120mg/po take one tablets once a day
Arm/Group | Control: Losartan / Week 12 -ITT | Test: Fimasartan / Week 12 -ITT
Number analyzed (Participants) | 238 | 247
mmHg | -8.56 (7.72) | -11.26 (7.53)
Statistical Analysis 1: Comparison: Control: Losartan / Week 12 -ITT vs Test: Fimasartan / Week 12 -ITT; Test type: Non-Inferiority — Non-Inferiority; p = 0.0001, t-test, 2 sided; Paired t-test

2. Secondary Outcome: Diastolic Blood Pressure Change
Description: * Value of DBP at 4 Weeks minus value of DBP at Baseline while in a sitting position
  * Value of DBP at 8 Weeks minus value of DBP at Baseline while in a sitting position
Time Frame: baseline and 4 weeks, 8 weeks
Population: As ITT group, these are subjects who have been randomly assigned and have at least one primary end point.
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Control: Losartan / Week 4,8 -ITT: Losartan group
  Losartan (Control): Losartan 50 mg ~ 100 mg/po, take one tablets once a day
- Test: Fimasartan / Week 4,8 -ITT: Fimasartan 60mg, 120mg
  Fimasartan: Fimasartan 60 ~ 120mg/po take one tablets once a day
Arm/Group | Control: Losartan / Week 4,8 -ITT | Test: Fimasartan / Week 4,8 -ITT
Number analyzed (Participants) | 238 | 247
mmHg
  Week 4 | -5.73 (6.56) | -8.22 (7.35)
  Week 8 | -8.01 (7.16) | -11.01 (7.63)
Statistical Analysis 1: Comparison: Control: Losartan / Week 4,8 -ITT vs Test: Fimasartan / Week 4,8 -ITT; Test type: Non-Inferiority — Non-Inferiority; p = 0.0001, t-test, 2 sided; Paired t-test

ADVERSE EVENTS:
Arm/Group | Control: Losartan | Test: Fimasartan
Serious Adverse Events (participants affected / at risk) | 5/250 | 3/255
Other Adverse Events (participants affected / at risk) | 76/250 | 82/255
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control: Losartan (N=250) | Test: Fimasartan (N=255)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
coronary artery occlusion (Cardiac disorders) | 1 (1) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Multiple fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control: Losartan (N=250) | Test: Fimasartan (N=255)
Headache (Nervous system disorders) | 17 (18) | 16 (17)
Dizziness (Nervous system disorders) | 9 (10) | 11 (11)
Hypoaesthesia (Nervous system disorders) | 2 (2) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 2 (2)
Dysaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Dysarthria (Nervous system disorders) | 1 (1) | 0 (0)
Global amnesia (Nervous system disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 5 (5) | 2 (2)
Nausea (Gastrointestinal disorders) | 4 (4) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1) | 3 (3)
Gastritis (Gastrointestinal disorders) | 4 (4) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dental caries (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis erosive (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Palatal oedema (Gastrointestinal disorders) | 0 (0) | 1 (1)
Tongue discolouration (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 5 (6) | 8 (8)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 5 (5)
Rhinitis (Infections and infestations) | 3 (3) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 1 (1) | 0 (0)
Otitis media acute (Infections and infestations) | 0 (0) | 1 (1)
pharyngitis (Infections and infestations) | 1 (1) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pelvic deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 4 (4)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 4 (4)
Blood urine present (Investigations) | 0 (0) | 2 (2)
Glucose urine present (Investigations) | 2 (2) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1)
Low density lipoprotein increased (Investigations) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 1 (1)
Spinal X-ray abnormal (Investigations) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 3 (3) | 3 (3)
Chest pain (General disorders) | 2 (2) | 2 (2)
Asthenia (General disorders) | 0 (0) | 2 (2)
Face oedema (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 4 (4)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Urticaria localised (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 2 (2) | 3 (3)
Tachycardia (Cardiac disorders) | 2 (2) | 0 (0)
Supraventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Blepharospasm (Eye disorders) | 1 (1) | 0 (0)
Conjunctivitis allergic (Eye disorders) | 0 (0) | 1 (1)
Eye pruritus (Eye disorders) | 0 (0) | 1 (1)
Eyelid ptosis (Eye disorders) | 1 (1) | 0 (0)
Keratoconjunctivitis sicca (Eye disorders) | 1 (1) | 0 (0)
Ocular hyperaemia (Eye disorders) | 0 (0) | 1 (1)
Xerophthalmia (Eye disorders) | 0 (0) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 2 (2) | 1 (1)
Eustachian tube dysfunction (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatitis alcoholic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal cyst (Renal and urinary disorders) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No